CLINICAL TRIAL: NCT06869512
Title: Cooperative Extension and Cancer Survivorship: Supportive Care Via Cooperative Extension Services (SUCCESS)
Brief Title: Cooperative Extension and Cancer Survivorship
Acronym: SUCCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17371
Record Dates: First submitted 2025-02-07; First posted 2025-03-11 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cancer Survivorship

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUCCESS Program (Experimental): This includes our cancer survivorship program which entails 6 weekly group education sessions. Each session includes 25 minutes of didactic and discussion-based lecture, 25 minutes of facilitated support group, and 10 minutes of brief group-based exercise.
  Interventions: Behavioral: SUCCESS

INTERVENTIONS:
Behavioral: SUCCESS — 6 group-based sessions with 25 minutes of didactic content, 25 minutes of facilitated support group, and 10 minutes of group physical activity

SUMMARY:
The goal of this clinical trial is to learn if a cancer survivor program, delivered via Cooperative Extension, is feasible and if it can improve health outcomes in cancer survivors who are post-active treatment.

Aim 1: Evaluate the feasibility and acceptability of SUCCESS. Hypothesis 1: SUCCESS will be feasible and acceptable as evidenced by delivery of the intervention among Educators (implementation), including in agreement with the curriculum in Phase 1 (fidelity) with >85% attendance (demand) among participants with >80% rating the intervention as acceptable or highly acceptable on 5-point Likert-type scale (acceptability).

Aim 2: Determine the preliminary efficacy of SUCCESS for improving HRQOL (primary outcome) and other psychosocial and health-related endpoints (e.g., financial toxicity) (secondary outcomes). Hypothesis 2: Compared to matched controls, adults LWBC who complete SUCCESS will have significant improvements in HRQOL per the PROMIS Global Health v1.2 at follow-up (i.e., after 6 weeks).

Aim 3: Examine changes in conserved transcriptional response to adversity (CTRA) gene expression in a subset of interventions participants at follow-up. Hypothesis 3: Adults LWBC who complete SUCCESS will experience significant CTRA down-regulation.

This is a single arm trial and there is no comparison group.

Participants will be asked to do survey- and Zoom-based data collection before and after completing the 6-week program.

ELIGIBILITY:
Inclusion Criteria:

* Previous adult-diagnosed cancer
* Post active cancer treatment
* No current active treatment, hormonal therapy permitted
* Ability to get to group sessions
* In Oklahoma

Exclusion Criteria:

* Current palliative or hospice care
* Surgical or medical history that precludes participation
* Positive screen on the Physical Activity Readiness Questionnaire+ (PAR-Q+) without a doctor's note approving study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delivery of sessions | Once per week for six weeks
  We will measure the percent of SUCCESS sessions delivered as planned by Educators
Fidelity to SUCCESS protocol | Once per week for six weeks
  We will measure what percentage of planned SUCCESS content is delivered as instructed.
Participant attendance | Once per week for six weeks
  We will measure how many enrolled participants attend each SUCCESS session
Acceptability of SUCCESS | Measured after SUCCESS (week 7-8 of the clinical trial)
  We will administer a feasibility survey after SUCCESS for participants to rate how much they liked it. Rating will be on a 5-point Likert Scale ("How would you rate this program?" 1=poor, 5=excellent)

SECONDARY OUTCOMES:
Diet quality | Baseline (week 1) and post-SUCCESS (week 7-8)
  We will measure diet quality as assessed via the National Cancer Institute Dietary Screener Questionnaire (DSQ). Outputs from the DSQ are intake of fruits and vegetables (cup equivalents), dairy (cup equivalents), added sugars (teaspoon equivalents), whole grains (ounce equivalents), fiber (g), and calcium (mg).
Physical function | Baseline (week 1) and post-SUCCESS (week 7-8)
  We will measure physical function using the 30-second Timed Chair Rise (30sTCR), measured in seconds.
Depressive symptoms | Baseline (week 1) and post-SUCCESS (week 7-8)
  Depressive symptoms will be measured using the Patient Health Questionnaire (PHQ-9). This provides a numeric score from 0-27, with higher=more depression
Anxiety symptoms | Baseline (week 1) and post-SUCCESS (week 7-8)
  Anxiety symptoms will be measured using the General Anxiety Disorder-7 (GAD-7). This provides a numeric score from 0-21, with higher=more anxiety.
Loneliness | Baseline (week 1) and post-SUCCESS (week 7-8)
  Loneliness will be measuring using the UCLA Loneliness Scale. This provides a numeric score from 20-80, with higher=more loneliness.
Social isolation | Baseline (week 1) and post-SUCCESS (week 7-8)
  Social isolation will be measured using the PROMIS Social Isolation Short Form (SF). This provides a numeric score from 4-20, with higher scores indicating more social isolation.
Financial Toxicity | Baseline (week 1) and post-SUCCESS (week 7-8)
  Financial toxicity will be measured using the COST: A FACIT Measure of Financial Toxicity (FACIT-COST). The FACT-COST provides a numeric score from 0-44, with higher meaning better financial well-being.
Health-related quality of life | Baseline (week 1) and post-SUCCESS (week 7-8)
  Health-related quality of life (HRQOL) will be measured using the PROMIS Global Health v1.2, which yields Global Physical Health and Global Mental Health Scores, both of which range numerically from 4-20; higher indicates better HRQOL.
Food insecurity | Baseline (week 1) and post-SUCCESS (week 7-8)
  Food insecurity will be measured using the USDA 6-item food insecurity screener. This yields a numeric score from 0-6, with higher=more food insecurity,
Basic psychological needs | Baseline (week 1) and post-SUCCESS (week 7-8)
  Basic psychological needs according to Self-Determination Theory (autonomy, competence, relatedness) will be measured using the Basic Psychological Need Satisfaction Scale. This provides three scores (one per psychological need) that ranges from 1-7, with higher=more of that need met.
Self-reported pain | Baseline (week 1) and post-SUCCESS (week 7-8)
  Pain will be measured using the Pain, Enjoyment, and General Activity (PEG) scale which provides a numeric score from 0-10, with 10=more pain and more interference from pain.
Conserved Transcriptional Response to Adversity (CTRA) gene expression | Baseline (week 1) and post-SUCCESS (week 7-8)
  Remote blood sampling procedures will be used to collect blood spots. RNA will be extracted from spots and sequenced for quantification of the 53-gene contrast score that comprises CTRA. This will only be done in a subset of participants.
Physical function | Baseline (week 1) and post-SUCCESS (week 7-8)
  We will measure physical function using 5 Times Sit-to-Stand (5xSTS) tests, measured in seconds.
Financial Toxicity | Baseline (week 1) and post-SUCCESS (week 7-8)
  Financial toxicity will be measured using the Composite Financial Burden Score (CFBS). The CFBS provides a numeric score from 0-6; higher scores denote increased financial burden.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Will be made available upon request.

REFERENCES:
- [Background] Pitasi O, Hildebrand D, Liebe R, Joyce J, Nagykaldi Z, Robertson MC, Braun A. Hiding in plain sight: Cooperative Extension as an underutilized approach to improving cancer survivorship outcomes in underserved populations. J Cancer Surviv. 2024 Oct 10. doi: 10.1007/s11764-024-01687-z. Online ahead of print. PMID 39388009